CLINICAL TRIAL: NCT06496750
Title: NIDA CTN-0132 Randomized, Double-Blind, Active Placebo-Controlled Trial of Ketamine for Methamphetamine Use Disorder (KMD)
Brief Title: Ketamine for Methamphetamine Use Disorder
Acronym: KMD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor-Psychiatry, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU-2023-1086
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorders; Substance Use; Methamphetamine Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Participants will receive IV ketamine (0.50mg/kg) dissolved in 0.9% sodium chloride in a total volume of 100mL and administered with an infusion pump at a constant rate over 40 minutes. IV ketamine will be administered 8 times over 6 weeks.
  Interventions: Drug: Ketamine Hydrochloride
- Midazolam (Active Comparator): Participants will receive IV midazolam (0.02mg/kg) dissolved in 0.9% sodium chloride in a total volume of 100mL and administered with an infusion pump at a constant rate over 40 minutes. IV midazolam will be administered 8 times over 6 weeks.
  Interventions: Drug: Midazolam Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Participants will receive IV ketamine (0.50mg/kg) dissolved in 0.9% sodium chloride in a total volume of 100mL and administered with an infusion pump over 45 minutes. Duration of each infusion may be extended by the Study Clinician supervising study medication infusion if slower infusion rate is better tolerated.
  Other Names: Ketelar
  Arms: Ketamine
Drug: Midazolam Hydrochloride — Participants will receive IV midazolam (0.02mg/kg) dissolved in 0.9% sodium chloride in a total volume of 100mL and administered with an infusion pump over 45 minutes. Duration of each infusion may be extended by the Study Clinician supervising study medication infusion if slower infusion rate is better tolerated.
  Other Names: Versed
  Arms: Midazolam

SUMMARY:
This study aims to determine whether treatment response with IV ketamine is superior to treatment response with IV midazolam in adults with moderate to severe MUD.

The study design is a 12-week randomized, double-blind, controlled trial comparing intravenous (IV) ketamine against IV midazolam, delivered over six weeks in 120 adults with moderate to severe methamphetamine use disorder (MUD).

DETAILED DESCRIPTION:
Effective management for methamphetamine use disorder (MUD) remains elusive, despite widespread misuse of this stimulant. Psychological interventions have demonstrated modest benefits, and relapse rates are high. There are currently no Food and Drug Administration (FDA)-approved pharmacotherapies for MUD. This study explores the efficacy, safety, and feasibility for intravenous (IV) ketamine as a treatment for MUD and will help to determine the effect size for a larger, multi-site trial of intravenous (IV) ketamine in MUD.

Participants will receive either IV ketamine (0.50mg/kg) or IV midazolam (0.02mg/kg) over 45 minutes per infusion for a total of eight (8) infusions over six (6) weeks. Medical management sessions with a study clinician will be provided to all participants once weekly (from Weeks 1 through 6).

The use of IV ketamine in this trial is consistent in dose (0.5 mg/kg) and duration of infusion (45-minute-long) to other studies of ketamine for psychiatric disorders (such as major depressive disorder and post-traumatic stress disorder, both of which are often comorbid in individuals with MUD) and substance use disorder. However, IV ketamine has not been directly evaluated as mono-pharmacotherapy in those with MUD yet.

Additionally, participants will be asked to participate in cognitive behavioral therapy (CBT) sessions once weekly (from Weeks 1 through 12) on a non-infusion day.

ELIGIBILITY:
Inclusion criteria

Study participants must:

1. Be 18 to 65 years old
2. Be able to sufficiently understand, speak, and read English
3. Be interested in reducing or stopping methamphetamine use
4. Meet criteria for methamphetamine use disorder
5. Use acceptable methods of contraception during participation in the study

Exclusion criteria

Study participants must not:

1. Have been in a research study of pharmacological or behavioral treatment for addiction within 6 months prior to written informed consent
2. Be currently in jail, prison, or inpatient overnight facility as required by court of law
3. Have upcoming surgery planned or scheduled
4. Be currently pregnant, breastfeeding, or planning on conception, if biologically female

Additional inclusion and exclusion criteria will be assessed by the study investigators at the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Treatment Response | 2 weeks
  Defined as having at least three methamphetamine-negative urine samples out of four samples obtained during Weeks 3 and 4.

SECONDARY OUTCOMES:
Non-serious adverse outcomes associated with IV ketamine treatment for methamphetamine use | 6 weeks
  Defined by non-serious adverse events (associated with the IV ketamine treatment) reported during the study intervention phase (weeks 1 to 6). Participants will be assessed for adverse events at each study visit.
Adherence to treatment | 6 weeks
  Defined by completion of at least five out of eight IV ketamine or IV midazolam infusions.
Total abstinence | 2 weeks
  Defined as four out of four methamphetamine-negative urine samples obtained during Weeks 3 and 4 (since missing urine drug screens will be counted as positive).
Abstinence from methamphetamine use | 12 weeks
  Defined by the self-reported days of methamphetamine use as reported on the Timeline Followback (TLFB) from Week 1 to Week 4, Week 5 to Week 6, and Week 7 to Week 12.
Differences in methamphetamine-negative urine samples from Weeks 1 to 6 and between ketamine and midazolam arms. | 6 weeks
  Urine samples will be collected twice a week at in-person visits.
Differences in methamphetamine-negative urine samples from Weeks 1 and 2 versus Weeks 3 and 4. | 4 weeks
  Urine samples will be collected twice a week at in-person visits.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Jha, MBBS, Principal Investigator — Associate Professor
Locations (4):
- United States (4):
  - Interdisciplinary Substance Use and Brain Injury Facility, Albuquerque, New Mexico
  - Addiction Institute of Mount Sinai, New York, New York
  - Prisma Health, Greenville, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No